CLINICAL TRIAL: NCT07284017
Title: The Impact of Neuronavigation in Repetitive Transcranial Magnetic Stimulation (rTMS) for Hemiplegic Stroke Patients.
Brief Title: The Impact of Neuronavigation in rTMS for Hemiplegic Stroke Patients.
Acronym: NeurorTMS-HS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Ting-Chun Fang, Attending Physician, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCVGH-CF25252C
Record Dates: First submitted 2025-11-30; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Hemiparesis After Stroke
Keywords: rTMS; Repetitive Transcranial Magnetic Stimulation; Neuronavigation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel assignment study where thirty participants with subacute stroke hemiparesis are randomly assigned to one of two groups for intervention. Both groups receive the identical low-frequency rTMS treatment, consisting of ten sessions of 1 Hz stimulation with 1,200 pulses per session, administered over two consecutive weeks. The primary distinction between the arms is the coil localization method: the Experimental Arm utilizes a neuronavigational system to guide and record the precise M1 hotspot positioning during each session, while the Control Arm relies on standard manual localization, such as cap positioning. The study is designed to compare the precision in coil placement and the resulting clinical efficacy of these two methods for motor recovery.
Who Masked: Participant
Masking Description: The study is single-blinded. Participants are masked to their group assignment (neuronavigation-guided rTMS versus conventional rTMS). Due to the inherent differences in the physical setup of the intervention, the personnel administering the rTMS treatment (Care Providers/Investigators) cannot be masked. However, the personnel responsible for evaluating the primary and secondary outcomes (Outcomes Assessors) will be masked to the participants' group assignment to ensure objective measurement of the Fugl-Meyer Assessment (FMA) and other clinical scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuronavigation-Guided Low-Frequency rTMS (Experimental): Participants in this arm receive low-frequency rTMS where the coil positioning is guided and recorded by a neuronavigational system during each of the 10 sessions. The system ensures precise targeting of the M1 hotspot contralateral to the lesion.
  Interventions: Device: Neuronavigation-Assisted rTMS for Stroke Hemiparesis
- Conventional Positioning Low-Frequency rTMS (Active Comparator): Participants in this arm receive the same low-frequency rTMS, but the coil positioning is performed via Standard Manual Localization (e.g., using cap positioning) over the M1 hotspot.
  Interventions: Device: Standard Localization rTMS for Stroke Hemiparesis

INTERVENTIONS:
Device: Neuronavigation-Assisted rTMS for Stroke Hemiparesis — Low-frequency (1 Hz) rTMS targeting the M1 "hotspot" contralateral to the lesion, delivered at 80% motor threshold (MT). Each session consists of 1,200 pulses (10 seconds ON, 1 second OFF, repeated 120 cycles). Treatment schedule: 1 session daily, 5 days/week, for 2 consecutive weeks (10 sessions total). Coil positioning is guided by a neuronavigational system using infrared camera and tracking balls.
  Arms: Neuronavigation-Guided Low-Frequency rTMS
Device: Standard Localization rTMS for Stroke Hemiparesis — Low-frequency (1 Hz) rTMS targeting the M1 "hotspot" contralateral to the lesion, delivered at 80% MT. Each session consists of 1,200 pulses (10 seconds ON, 1 second OFF, repeated 120 cycles). Treatment schedule: 1 session daily, 5 days/week, for 2 consecutive weeks (10 sessions total). Coil positioning is performed using standard manual localization with cap positioning.
  Arms: Conventional Positioning Low-Frequency rTMS

SUMMARY:
This is a randomized, controlled trial investigating the efficacy and precision of neuronavigation -guided repetitive transcranial magnetic stimulation (rTMS) for motor recovery in patients with subacute stroke hemiparesis.

The primary goal is to determine if using neuronavigation to precisely target the unaffected primary motor cortex (M1) improves treatment accuracy, efficiency, and clinical outcomes compared to conventional manual positioning.

The study will enroll 30 participants with first-ever stroke onset between 2 weeks and 6 months. Participants will be randomized into two parallel groups: the Experimental Group (neuronavigation-guided rTMS) and the Control Group (conventional positioning rTMS). Both groups will receive the same rTMS parameters: 1 Hz stimulation (low-frequency) over the unaffected M1, 1,200 pulses per session, administered for 10 sessions over 2 consecutive weeks.

Primary outcome measures include the change in the Fugl-Meyer Assessment (FMA) Score for the Upper Extremity and the measurement of coil positioning deviation between sessions. Assessments will be conducted at baseline (T0), post-treatment (T1, Week 3), and one month post-treatment (T2, Week 7). This study is funded in part by a research grant from the Metal Industries Research & Development Centre (MIRDC).

DETAILED DESCRIPTION:
This is a single-center, randomized, two-group parallel-assignment interventional trial conducted at Taichung Veterans General Hospital to compare the effectiveness of neuronavigation-guided rTMS versus conventional rTMS in subacute stroke patients with hemiparesis.

Background: Repetitive Transcranial Magnetic Stimulation (rTMS) is recognized for its potential in stroke rehabilitation, with low-frequency (1 Hz) stimulation over the unaffected motor cortex in the subacute phase rated as Grade A (definitely effective) for upper limb motor recovery. However, the efficacy of rTMS is highly dependent on accurate and consistent coil placement over the target cortical area.

Study Hypothesis: We hypothesize that using neuronavigation-which integrates infrared tracking with brain MRI to establish a precise 3D coordinate reference-will significantly increase the treatment precision, reduce the required localization time, and ultimately lead to superior clinical outcomes compared to conventional manual targeting methods.

Intervention Details:

1. Participants: 30 eligible patients (age 20-85) who are 2 weeks to 6 months post-stroke and demonstrate unilateral upper limb weakness will be enrolled.
2. Stimulation Parameters: All participants will receive low-frequency rTMS (1 Hz) at 80% of the motor threshold (RMT). Each session consists of 1,200 pulses delivered over approximately 20 minutes.
3. Grouping:

(1)Experimental Group (n=15): Coil positioning will be guided by a neuronavigational system throughout all 10 sessions. The system tracks the coil and patient's head relative to the initial M1 hotspot.

(2)Control Group (n=15): Coil positioning will rely on standard manual localization (e.g., cap positioning).

Outcome Assessments:

The study will track three primary outcomes: FMA score (a key measure of motor function), coil positioning deviation (a measure of precision), and the time required for initial hotspot localization. Secondary outcomes include functional and spasticity measures such as the Barthel Index (BI), Modified Rankin Scale (mRS), Modified Ashworth Scale (mAS), and neurophysiological parameters (MEP, EEG).

Timeline:

All outcome measures will be assessed at three time points: Baseline (T0), Post-treatment (T1, Week 3), and 1-month Follow-up (T2, Week 7).

Safety:

All adverse events, including rare severe events like seizures (<0.01%) and syncope, will be managed according to standard emergency protocols, and treatment will be discontinued if adverse effects persist or significant clinical weakness occurs. The study protocol is within established safety guidelines.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic or hemorrhagic stroke confirmed by imaging.
* Stroke causing unilateral upper limb weakness (MRC grade <=3)
* Stroke onset must be between 2 weeks and 6 months prior to enrollment (subacute phase).
* Age between 20 and 85 years old.
* Stable vital signs, clear consciousness, and no cognitive impairment.
* Able to cooperate with assessments and treatment.
* Written informed consent must be signed by the patient or a legal guardian.

Exclusion Criteria:

* Contraindications to TMS (e.g., metallic implants in head, pacemaker, cochlear implant).
* History of epilepsy or seizures.
* Pregnancy.
* Severe cognitive or communication disorders, or inability to give informed consent.
* Unstable medical conditions affecting participation.
* Use of certain medications, including benzodiazepines, antidepressants, muscle relaxants (baclofen, tizanidine), or ongoing botulinum toxin injections for post-stroke spasticity.
* Modified Rankin Scale (mRS) score >=5 .

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) Score | Baseline (T0), Post-treatment (T1, 2 weeks), and 1 Month Post-treatment (T2)
  The FMA is a quantitative, reliable, and widely used stroke-specific assessment tool for measuring motor recovery. This scale ranges from 0 to 66 points, where a higher score indicates better motor function of the upper limb. The difference in FMA scores between the neuronavigation group and the standard localization group will be compared to evaluate the treatment efficacy.
Deviation in Coil Positioning | Intra-session (recorded during each daily treatment session for 2 weeks) and Inter-session (change from baseline to 2 weeks)
  This measure quantifies the positional stability and accuracy of the rTMS coil placement. The neuronavigational system records positional coordinates before and after each session in the experimental group. The outcome will compare the intra-session (stability throughout a single treatment) and inter-session (change from baseline to 2 weeks) deviation in coil coordinates between the neuronavigation-guided group and the standard manual localization group.
Time Required for Initial Hotspot Localization | Baseline (T0)
  This outcome measures the time (recorded in seconds or minutes) needed to accurately determine the M1 "hotspot" (the site eliciting the maximal motor-evoked potential (MEP)) at the start of the study. This comparison aims to quantify the efficiency difference between the neuronavigation-guided method and the standard manual localization method.